CLINICAL TRIAL: NCT06654596
Title: A Multicenter, Randomized, Controlled Clinical Study on the Efficacy and Safety of Telitacicept in Patients with IgA Nephropathy
Brief Title: Efficacy and Safety of Telitacicept in IgAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); RenJi Hospital (Other); Sichuan Provincial People's Hospital (Other); Renmin Hospital of Wuhan University (Other); Shanghai 6th People's Hospital (Other); Shanghai Longhua Hospital (Unknown); Huashan Hospital (Other); Shanghai Changzheng Hospital (Other); Wannan Medical College Yijishan Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Songjiang Hospital Affiliated to Shanghai Jiaotong University School of Medicine (Other Government)
Responsible Party: Principal Investigator, Xie Jingyuan, MD, Chief physician, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TETA-IgA
Record Dates: First submitted 2024-10-18; First posted 2024-10-23 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: IgA Nephropathy (IgAN); Kidney Diseases; Telitacicept; Glucocorticoid
MeSH Terms: conditions — Glomerulonephritis, IGA; Kidney Diseases | interventions — telitacicept; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telitacicept+ACEI/ARB (Experimental)
  Interventions: Drug: Telitacicept 240mg
- Glucocorticoids+ACEI/ARB (Active Comparator)
  Interventions: Drug: Glucocorticoid

INTERVENTIONS:
Drug: Telitacicept 240mg — Patients in telitacicept group will be treated with maximum tolerable dose of angiotensin converting enzyme inhibitor ( ACEI ) and/or angiotensin II receptor blocker ( ARB ) combined with telitacicept. 240 mg telitacicept will be used once a week for 40 weeks.
  Arms: Telitacicept+ACEI/ARB
Drug: Glucocorticoid — Patients in glucocorticoid group will be treated with ACEI/ARB and glucocorticoid ( prednisone/prednisolone) 0.5mg/kg (maximum 40mg/d). After 8 weeks, reduce the dosage by 5 mg per month for a total of 28-40 weeks.
  Arms: Glucocorticoids+ACEI/ARB

SUMMARY:
A study to evaluate efficacy and safety of telitacicept in the treatment of patients with primary IgA nephropathy at high risk of progression.

DETAILED DESCRIPTION:
IgA nephropathy is a glomerulonephritis characterized by pathological IgA deposition in the mesangial region. Its clinical and pathological manifestations are diverse and heterogeneous. Its pathogenesis has not yet been fully clarified, and there is currently no unified treatment plan. As a recombinant human B lymphocyte stimulator receptor-antibody fusion protein, telitacicept has become a new therapeutic target. The results of the Phase II clinical trial of this drug for IgA nephropathy have already been published. It is one of the key pioneering clinical studies in the field of IgA nephropathy treatment. The study showed that telitacicept can effectively reduce patients' proteinuria and reduce the risk of disease progression. Based on the above research results, the investigators plan to conduct a multicenter, randomized, controlled clinical study to evaluate the efficacy and safety of telitacicept in the treatment of primary IgA nephropathy patients with a high risk of progression.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old, male or female
2. Primary IgA nephropathy confirmed by renal biopsy.
3. Urine protein ≥ 0.75g/24h or 24-hour urine protein creatinine ratio (PCR) ≥ 0.6 g/g.
4. eGFR ≥ 25 ml/min/1.73 m2 calculated using the CKD-EPI formula.
5. Received treatment with ACEI/ARB for 12 weeks before randomization, and the drug dose (within the maximum tolerated range) was stable within 4 weeks before randomization.
6. Use of SGLT2, MRA, hydroxychloroquine, and etc. remained unchanged.
7. Voluntarily participated in this study and signed the informed consent form.

Exclusion Criteria:

1. Patients with abnormal laboratory indicators (see study protocol for details).
2. Secondary IgA nephropathy such as Henoch-Schonlein purpura, SLE, cirrhosis, etc.
3. Use of systemic glucocorticoids/immunosuppressants within 3 months (such as cyclophosphamide, azathioprine, mycophenolate mofetil, leflunomide, tacrolimus, cyclosporine, tripterygium wilfordii, etc.).
4. Use of biological agents within 6 months (rituximab, etc.).
5. Active infection, such as active tuberculosis, active hepatitis, hepatitis C, herpes zoster, HIV, etc. According to the results of the five hepatitis B test: patients with positive HBsAg should be excluded; patients with negative HBsAg but positive HBcAb, regardless of whether HBsAb is positive or negative, need to test HBV-DNA to determine their situation: if HBV-DNA is positive, the patient needs to be excluded; if HBV-DNA is negative, the patient can participate in the trial.
6. COVID-19 infection within 2 weeks before randomization.
7. Live vaccine within 4 weeks before randomization.
8. History of malignant tumor within five years.
9. Uncontrolled hypertension (systolic blood pressure>140mmHg or diastolic blood pressure>90mmHg).
10. Poorly controlled diabetes (glycosylated hemoglobin>8%).
11. Pregnant women and breastfeeding women.
12. Participating in other clinical trials at the same time.
13. Surgery, chemotherapy, radiotherapy and other treatments are planned during the study.
14. Other reasons judged by researchers as unsuitable for inclusion in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change of 24-hour urine protein | From baseline to week 40
  Change of 24-hour urine protein from baseline to week 40

SECONDARY OUTCOMES:
Change of PCR | From baseline to week 40
  Change of 24-hour urine protein creatinine ratio (PCR) from baseline to week 40
Annualized eGFR slope | From baseline to week 40
  Annualized eGFR slope from baseline to week 40
Change of eGFR | From baseline to week 40
  Change of eGFR from baseline to week 40
Proportion of patients with a decrease in eGFR ≥30% | From baseline to week 40
  Proportion of patients with a decrease in eGFR ≥30% from baseline to week 40
Proportion of patients with a decrease in eGFR ≥40% | From baseline to week 40
  Proportion of patients with a decrease in eGFR ≥40% from baseline to week 40
Change of 24-hour urine ACR | From baseline to week 40
  Change of 24-hour urine albumin creatinine ratio (ACR) from baseline to week 40
Proportion of patients achieving 24-hour urine PCR < 0.6 g/g | From baseline to week 40
  Proportion of patients achieving 24-hour urine PCR < 0.6 g/g from baseline to week 40
Time from the first use of treatment to the occurrence of a composite endpoint event | Up to 40 weeks
  Time from the first use of treatment to the occurrence of a composite endpoint event. The composite endpoint event was defined as: the time from the first use of treatment to the first decrease in eGFR from baseline by ≥30% or ≥40% (at least 4 weeks), initiation of maintenance renal dialysis (at least 4 weeks), eGFR <15 mL/min/1.73m2 (at least 4 weeks), renal transplantation, or death due to renal failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, China